CLINICAL TRIAL: NCT04210102
Title: Accuracy of Lung Ultrasound for the Diagnosis of Community-Acquired Pneumonia in Emergency Room Patients
Brief Title: Community-Acquired Pneumonia Diagnosis Using Lung Ultrasound in Emergency Room Adults
Acronym: CAPUERA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-14
Record Dates: First submitted 2019-12-11; First posted 2019-12-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: Prospective and randomised study in 2 parallel groups to compare diagnosis performance of LUS and CR as a primary imaging for diagnosis of CAP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR + LUS (Other): Patient will be performed first the Chest radiography then the Lung ultrasound.
  Interventions: Diagnostic Test: Lung Ultrasound (LUS); Diagnostic Test: Chest radiography (CR)
- LUS + CR (Other): Patient will be performed first the Lung ultrasound then the Chest radiography
  Interventions: Diagnostic Test: Lung Ultrasound (LUS); Diagnostic Test: Chest radiography (CR)

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound (LUS) — Lung Ultrasound : Ultrasound is a medical imaging technique that relies on the use of ultrasound, inaudible sound waves, which allow to "visualize" lungs.
Diagnostic Test: Chest radiography (CR) — The chest X-ray is a medical imaging examination that provides images of the lungs through the X-ray pulse.

SUMMARY:
Community-Acquired Pneumonia (CAP) is a major problem in Emergency Department (ED). Diagnosis relies on combination of clinical symptoms and results of chest radiography (CR). Patients' management (treatment, support) depends on delay and quality of the diagnosis. However, signs and symptoms are highly aspecific and interpretation of CR is subject to frequent discrepancies. Then diagnosis of CAP may be uncertain; therefore, overdiagnosis is frequent and leads to over-use of antimicrobial therapy; missing diagnosis is also deleterious and delays adequate treatment including antibiotics. CT scan completes CR and helps clinician making properly diagnosis of CAP; obtaining CT in a 4-hour time-lapse allows better diagnosis and management as accurate as an independent expert adjudication committee does. However availability of CT as well as radiation interrogates on the benefit that Lung Ultrasounds (LUS) may have in diagnosis strategy of suspected CAP. LUS is a noninvasive easy-to-use device whose practice is widely endorsed worldwide by emergency medicine associations and societies. Additionally, previous studies advocate for the use of LUS for diagnosis of CAP in the ED. Therefore the Promotor developed a study to compare LUS and CR as a primary imaging for diagnosis of CAP at the ED.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+)
* Suspected CAP by attending emergency physician
* And new onset of systemic infection (at least one among sweat, chills, aches and pain, temperature ≥38°C or <36°C)
* And symptoms of an acute lower respiratory tract infection (at least one among cough, sputum production, dyspnea, chest pain, altered breathing sounds at auscultation
* No previous imaging for the current medical problem
* Inform consent (signed)
* Affiliation to insurance (France, Monaco)

Exclusion Criteria:

* Age below 18-year of age
* Patients in palliative care
* Pregnant women
* anticipated barriers to completing follow-up data collection,
* patients classified three or higher according to the CRB65 score,
* patients requiring intensive care for any purpose because of specific management of critically ill
* refusal to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of lung ultrasound (LUS) and chest X-ray (CR) to detect community-acquired pneumonia (CAP) will be mesured and compared in patients visiting the emergency department for suspected CAP | Within the day of inclusion

SECONDARY OUTCOMES:
specificity, positive predictive value and negative predictive value : indicators of diagnosis performance, will be measured and compared as a primary imaging for diagnosis of CAP | Within the day of inclusion
Specificity, positive predictive value, negative predictive value will be measured and compared in each sequence of imaging (CR + LUS and LUS + CR) for CAP detection | Within the day of inclusion
medical decisions for diagnosis of CAP after each step LUS then CR or CR then LUS and after low dose CT6scan (CT) will be compared to the medical decisions of the adjudication committee | Up to 6 months
The concordance of interpretation (for CR and CT) between attending radiologist and expert radiologist of the adjudication committee (gold standard) wil be studied. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: CLAESSENS Yann-Erick, MD, PhD, Principal Investigator — CH Princesse Grâce
Locations (1):
- CHPG, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorca J, Torres A. Lower respiratory tract infections in the community: towards a more rational approach. Eur Respir J. 1996 Aug;9(8):1588-9. doi: 10.1183/09031936.96.09081588. No abstract available. PMID 8866576
- [Background] Woodhead M. Community-acquired pneumonia in Europe: causative pathogens and resistance patterns. Eur Respir J Suppl. 2002 Jul;36:20s-27s. doi: 10.1183/09031936.02.00702002. PMID 12168744
- [Background] Claessens YE, Debray MP, Tubach F, Brun AL, Rammaert B, Hausfater P, Naccache JM, Ray P, Choquet C, Carette MF, Mayaud C, Leport C, Duval X. Early Chest Computed Tomography Scan to Assist Diagnosis and Guide Treatment Decision for Suspected Community-acquired Pneumonia. Am J Respir Crit Care Med. 2015 Oct 15;192(8):974-82. doi: 10.1164/rccm.201501-0017OC. PMID 26168322